CLINICAL TRIAL: NCT02866981
Title: Observation for Patients With Asymptomatic CNS Metastatic Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-180EX
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Cancer; Metastatic Cancer
Keywords: Brain Metastases
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Brain Neoplasms | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Observation (Experimental): Patients that meet all inclusion and exclusion criteria are monitored every 2 months for two years or until a therapeutic intervention is warranted.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
The purpose of this registry is to determine if select patients with CNS metastatic disease can be safely observed rather than treated. The investigators hypothesize that there is a subset of patients with small asymptomatic CNS mets that do not require treatment, these patients can simply be observed and will not have CNS progression.

DETAILED DESCRIPTION:
Subjects will be given a consultation with physician investigators in the department of one of the study investigators, who will introduce the study if the subject is potentially eligible.

Information collected at initial assessment:

* Quality of life survey (FACT-Br)
* History and Physical exam (to include KPS, disease status on most recent non-CNS imaging, chemotherapy history, age).
* Measurement of walking pace: patient will walk a pre- measured 6 meters, patient is to be instructed to walk at a normal pace. The time required to travel this distance will be recorded. For patients that are wheelchair bound or otherwise immobile, the pace will be recorded as '0'.
* Neurocognitive testing (Montreal Cognitive Assessment)
* MRI scan with contrast (must be within 6 weeks)

Observation and Follow-up Visits:

* Patients will be seen at 6 weeks and then every 2 months for follow-up (with physical exam) with repeat MRI with contrast at that time
* FACT-Br survey to be filled out at each follow-up
* Neurocognitive status (Montreal Cognitive Assessment)

Treatment for Progression:

* Progression is defined as: Increase in size to > 1 cm (> 2.0 for patients being treated with targeted therapy); Interval growth of 0.4 cm in 6-8 weeks; Development of edema or increase in edema; Development of symptoms from CNS lesion; Patient preference
* Patients that meet criteria for treatment will be treated at discretion of treating physician; options can include whole brain radiation, radiosurgery, surgery.

The study does not provide financial or other compensation to subjects

ELIGIBILITY:
Inclusion Criteria:

* CNS metastatic disease that meets the following:
* No lesion greater than 0.8 cm for patients not on targeted therapy with CNS penetration
* No lesion greater than 1.5 cm for patients on targeted therapy with CNS penetration.
* No previous treatment for the observed lesion. Patients may have had other lesions that have been treated as long as there is at least one index lesion that has not been treated. For example, patient may have had 3 lesions treated in March 2012 with radiosurgery and on recent scan is found to have a new 0.5 cm lesion, this patient is eligible.
* Less than 5 untreated CNS lesions.
* Able to have MRI scan with contrast
* All CNS lesions are asymptomatic. Patient may have symptoms from previous treatment or cancer outside the CNS but cannot have symptoms attributable to the current CNS metastatic disease. This is left to the discretion of the treating physician and in some instances is not easy as sometimes CNS metastatic disease is incidental finding to un-related symptoms.
* Eligible primaries
* Lung (NSCLC)
* Lung (SCLC) that have had previous Whole brain radiation
* GI
* Head and Neck
* Gyn
* Prostate
* Breast
* Kidney
* Melanoma
* Sarcoma

Exclusion Criteria:

* CNS lesion that does not meet following:
* No lesion greater than 0.8 cm for patients not on targeted therapy with CNS penetration
* No lesion greater than 1.5 cm for patients on targeted therapy with CNS penetration.
* More than 5 CNS lesions (can have had previously treated lesions by either surgery or radiation, but at time of protocol SRS must have 5 or less untreated lesions).
* Symptomatic CNS lesions
* Ineligible primaries
* Lymphoma
* Primary CNS tumors
* SCLC that has not had previous whole brain radiation
* Leptomeningeal disease in CNS
* Patients unable to have an MRI (secondary for example to metal hardware)
* Patients unable to have MRI contrast (secondary for example to poor renal function
* CNS lesion >0.8 cm in any dimension for patients not on targeted therapy with CNS penetration or >1.5 cm for patients on targeted therapy with CNS penetration.
* Note that there is no KPS cut-off for eligibility

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-02; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Every two months for two years
  Kaplan-Meier survival analyses
CNS treatment-free survival rate | Every two months for two years
  overall survival combined with CNS treatment

SECONDARY OUTCOMES:
Quality of life | Every two months for two years
  determined by FACT-Br
Natural History of untreated CNS met | Every two months for two years
  Measure the size of CNS target lesion over time
Type of treatment | Every two months for two years
  When/if needed
Indication for treatment | Every two months for two years
  when/if treatment is needed due to discontinuation of observation. Classified between: increase in size to >1cm; interval growth of 0.4 cm in 6-8 weeks; development of edema or increase in edema; development of symptoms; or patient preference.
Neurocognitive testing | Every two months for two years
  Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Harry Mazurek, MD, Study Director — Cooper University Health System; Gregory Kubicek, MD, Principal Investigator — Cooper University Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No